CLINICAL TRIAL: NCT04409483
Title: Evaluation of Additional Treatments for COVID-19: a Randomized Trial in Niger
Acronym: TRASCOV
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Epidemic dynamics
Sponsor: Epicentre (Other)
Collaborators: Université Abdou Moumouni (Unknown); Centre de Recherche Médicale et Sanitaire (Other); Ministry of Public Health, Republic of Niger (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trascov
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — lopinavir-ritonavir drug combination; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Standard care for COVID-19 according to the national guidelines of Niger
  Interventions: Combination Product: Standard Care
- Standard Care plus lopinavir/ritonavir (Experimental): Standard care for COVID-19 according to the national guidelines of Niger plus lopinavir/ritonavir
  Interventions: Drug: Lopinavir-Ritonavir Drug Combination; Combination Product: Standard Care

INTERVENTIONS:
Drug: Lopinavir-Ritonavir Drug Combination — 400mg/100mg taken orally twice daily for 14 days.
  Arms: Standard Care plus lopinavir/ritonavir
Combination Product: Standard Care — Paracetamol as needed for the symptomatic treatment of fever and vitamin C 1000 mg daily

SUMMARY:
The purpose of this study is to assess whether lopinavir/ritonavir (or eventually other antiviral drugs) is effective at reducing the rate of hospitalization among confirmed COVID-19 cases treated as outpatients.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients who meet all eligibility criteria and who give written informed consent will be randomized to receive standard care or standard care plus lopinavir/ritonavir (400mg/100mg twice daily for 14 days). Participants will receive daily visits from study staff for 15 days and be followed for a total of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Suspect, probable or confirmed case of COVID-19
* Men and women aged ≥12 years, including pregnant and breastfeeding women
* SpO2 ≥93% on room air
* Signature of informed consent form

Exclusion Criteria:

* Medical indication for hospitalization at the time of enrolment
* Severe chronic liver disease
* Known infection with HIV
* Known allergy or severe intolerance to lopinavir/ritonavir
* Absolute contra-indication to lopinavir/ritonavir, including concomitant therapy with a medication whose metabolism is dependent on isoform CPY3A with a narrow therapeutic window (e.g., amiodarone, colchicine, simvastatin, lovastatin, etc.)
* Treatment with an antiviral medication in the 28 days prior to enrolment
* Dementia or other condition that interferes with active participation in data collection and obtaining informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization or death | 15 days following randomization
  Hospitalization associated with desaturation (SpO2 ≤92%) or death due to any cause

SECONDARY OUTCOMES:
All-cause mortality | 15 days following randomization
  Death due to any cause
All-cause mortality | 28 days following randomization
  Death due to any cause
Time to hospitalization | 28 days following randomization
  Length of time between randomization and hospitalization associated with desaturation (SpO2 ≤92%)
Length of hospitalization | 28 days following randomization
  Total duration of hospitalization associated with desaturation (SpO2 ≤92%)
Admission to intensive care | 28 days following randomization
  Proportion of participants admitted to an intensive care unit
Adverse events | 28 days following randomization
  Proportion of participants having an adverse event
Serious adverse events | 28 days following randomization
  Proportion of participants having a serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca F Grais, Study Director — Epicentre; Eric Adehossi, Principal Investigator — Hôpital Général de Référence de Niamey

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be shared with local and international authorities.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become fully accessible after primary publication of results.